CLINICAL TRIAL: NCT05539469
Title: A 6-months Evaluation of Patients' Compliance and Oral Hygiene During Rapid Maxillary Expander (RME) Treatment Using "Ortodontika" Smartphone Application: a Randomized Clinical Trial
Brief Title: A 6-months Evaluation of Patients' Compliance and Oral Hygiene During Rapid Maxillary Expander (RME) Treatment Using "Ortodontika" Smartphone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022-ORTODONTIKA
Record Dates: First submitted 2022-09-07; First posted 2022-09-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Maxillary Transverse Deficiency
Keywords: Oral hygiene; Rapid Maxillary Expander; Smartphone application; Orthopedic treatment

STUDY DESIGN:
Intervention Model Description: Two parallel arms.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): Patients from this group will be assisted by Orthodontika application during orthopedic treatment. Reminders will be sent for the activation of Rapid Maxillary Expander and for oral hygiene maneuvers. Written information about orthopedic treatment and oral hygiene tips can be read.
  Interventions: Device: Ortodontika app
- Control group (Other): Patients from this group will not have access to Orthodontika application during orthopedic treatment. Patients will receive only verbal instruction about the activation of Rapid Maxillary Expander and for oral hygiene maneuvers.
  Interventions: Other: Verbal instructions

INTERVENTIONS:
Device: Ortodontika app — parents will download and use Ortodontika smartphone application for all the duration of the study. It will be an aid during orthopedic treatment. During the activations, a notification will be set to remind the daily activation of RME. After the end of the activation protocol, parents will receive a notification every 2 weeks to instruct their children to proper oral hygiene maneuvers. Parents will have to show their children the videos for oral hygiene maintenance every 2 weeks until the end of the study.
  Arms: Trial group
Other: Verbal instructions — verbal instructions will be given chairside to patients and parents regarding RME activation and its cleaning, together with instructions for daily oral hygiene manoeuvres.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the clinical use of the smartphone application "Ortodontika" for the compliance of orthodontic patients with Rapid Maxillary Expander (RME).

Patients and parents consenting to participate in the study will sign the informed consent for their child. At the baseline (T0), a periodontal examination will be carried out by means of a probe assessing Bleeding Index, Plaque Index and Modified Gingival Index on upper first incisors, first premolars/first primary molars and first molars. A professional oral hygiene will be performed using a piezoelectric instrument and a manual scaler. A RME will be cemented with a glass ionomer cement on the maxillary first molars and will be activated by parents on clinicians' instructions. Patients will receive an oral hygiene kit containing toothpaste, soft-bristled toothbrush, single tufted brush and interdental brushes (0.6 and 0.9 mm). Orthodontic wax and 1% chlorhexidine will be given for emergencies. At this point, patients will be divided into two groups:

* Control group: verbal instructions on the correct activation of the RME and on its cleaning will be given to parents at each visit, together with verbal instructions on the correct daily practices for oral hygiene;
* Trial group: use of "Ortodontika" smartphone application as adjunct to verbal instructions on the correct activation of the RME to be performed by one parent, through a daily notification until T1 (end of activations); parents have to supervise daily oral hygiene of RME and the correct daily practices for oral hygiene. A notification will be sent every 2 weeks until the end of the study to remind patients to watch the videos on oral hygiene maneuverers.

Patients will be visited at the end the activations (T1), after 1.5 months (T2), after 3 (T3) and 6 months (T6). At the recall, the periodontal indices will be evaluated again. At each recall, extra products will be given for home oral hygiene Patients and parents from the Control group will receive a questionnaire to evaluate awareness of orthodontic therapy (aims and phases) and knowledge of oral hygiene maneuverers. Patients and parents from the Trial group will receive an extra questionnaire about Ortodontika application. During the study, the number of emergencies will be recorded.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical use of the smartphone application "Ortodontika" for the compliance of orthodontic patients with Rapid Maxillary Expander (RME).

Patients and parents consenting to participate in the study will sign the informed consent for their child. At the baseline (T0), a periodontal examination will be carried out by means of a probe (UNC probe 15; Hu-Friedy, Chicago, IL, USA) assessing Bleeding Index, Plaque Index and Modified Gingival Index on upper first incisors, first premolars/first primary molars and first molars. A professional oral hygiene will be performed using a piezoelectric instrument (Multipiezo, Mectron S.p.a, Carasco, Italy) and a manual scaler (LM23, LM-Dental, Pargas, Finland). A RME will be cemented with a glass ionomer cement (3M Multi-Cure, 3M Unitek, Monrovia, CA, USA) on the maxillary first molars and will be activated by parents on clinicians' instructions. Patients will receive an oral hygiene kit containing toothpaste (GUM Junior 7+, Sunstar Deutschland GmbH, Schonau, Germany), soft-bristled toothbrush (GUM Technique PRO toothbrush), interdental brush 0.6 and 0.8 mm of diameter (GUM TRAV-LER) and a single tufted brush (GUM End-Tuft). Orthodontic wax will be given for emergencies related to RME (GUM ORTHO wax) and 1% chlorhexidine gel (Curasept Periodontal gel, Curasept S.p.A, Saronno, VA, Italy) will be given for gingival inflammation. At this point, patients will be divided into two groups:

* Control group: verbal instructions on the correct activation of the RME and on its cleaning will be given to parents at each visit, together with verbal instructions on the correct daily practices for oral hygiene;
* Trial group: use of "Ortodontika" smartphone application as adjunct to verbal instructions on the correct activation of the RME to be performed by one parent, through a daily notification until T1 (end of activations); parents will have to supervise daily oral hygiene of RME and the correct daily practices for oral hygiene. A notification will be sent every 2 weeks until the end of the study to remind patients to watch the videos on oral hygiene maneuverers.

Patients will be visited at the end of the activations (T1), after 1.5 months (T2), after 3 (T3) and 6 months (T6). At the recall, the periodontal indices will be evaluated and a questionnaire will be given to patients. At each recall, extra products will be given for home oral hygiene. During the study, the number of emergencies will be recorded: RME decementation, patients perceiving pain related to plaque accumulation, mucosal ulcerations due to vestibular tubes, parents that do not understand how to perform RME activations, patients asking the clinician to perform RME activations chairside. A questionnaire will be given to patients and parents belonging to both groups to evaluate awareness of orthodontic therapy aims and phases, knowledge of oral hygiene maneuverers. A questionnaire about Ortodontika application usefulness will be given only to patients and parents belonging to Trial group.

ELIGIBILITY:
Inclusion Criteria:

* patients and their parents are able or willing to give informed consent;
* patients who will begin orthopedic treatment with RME cemented on first maxillary molars and with welded vestibular tubes;
* patients undergone no previous orthopedic/orthodontic treatment;
* parents' willing to download and use Ortodontika application;
* parents possessing an Apple or Android smartphone with iOS ≥ 10.0 or Android ≥ 4.4 versions;
* smartphone provided with an internet connection.

Exclusion Criteria:

* no sectional wire appliances in the upper arches;
* no need of additional orthopedic/orthodontic appliances, also in the lower arch;
* no vestibular welded protraction hooks on RME;
* patients taking regular medications for systemic diseases that could alter periodontal conditions and pain perception (antibiotics, antibacterial mouth rinses, NSAIDS, steroids);
* siblings with previous orthopedic treatment with RME;
* parents and patients with low compliance.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Change in Modified Gingival Index (Eppright et al., 2014) | Baseline (T0), 1 month (end of activations - T1), after 1.5 months (T2), after 3 (T3) and 6 months (T6)
  Scoring criteria (one measurement for each tooth: upper first incisors, first premolars/first primary molars and first molars):
  0. Absence of inflammation
  1. Mild inflammation (marginal or papillary unit)
  2. Mild inflammation (entire marginal and papillary unit)
  3. Moderate inflammation
  4. Severe inflammation
Change in Bleeding Index (Saxton and van der Ouderaa, 1989) | Baseline (T0), 1 month (end of activations - T1), after 1.5 months (T2), after 3 (T3) and 6 months (T6)
  Scoring criteria (mesio-buccal, direct buccal, and disto-buccal probed gingival sulci of upper first incisors, first premolars/first primary molars and first molars):
  0. Absence of bleeding after 30 seconds
  1. Bleeding observed after 30 seconds
  2. Immediate bleeding
Change in Plaque Index (Quigley et al. 1962) | Baseline (T0), 1 month (end of activations - T1), after 1.5 months (T2), after 3 (T3) and 6 months (T6)
  Scoring criteria (one measurement for the buccal surface of upper first incisors, first premolars/first primary molars and first molars):
  0. No plaque
  1. Discontinuous band of plaque at gingival margin
  2. Up to 1-mm continuous band of plaque at gingival margin
  3. Band of plaque wider than 1 mm but less than 1/3 of surface
  4. Plaque covering between 1/3 and 2/3 of surface
  5. Plaque covering 2/3 or more of surface
Change in Number of emergencies | Baseline (T0), 1 month (end of activations - T1), after 1.5 months (T2), after 3 (T3) and 6 months (T6)
  RME decementation, patients perceiving pain related to plaque accumulation, mucosal ulcerations due to vestibular tubes, parents that do not understand how to perform RME activations, patients asking the clinician to perform RME activations chairside will be collected.
Change in Awareness questionnaire | Baseline (T0), 1 month (end of activations - T1), after 1.5 months (T2), after 3 (T3) and 6 months (T6)
  Parents and patients from both the groups will complete a questionnaire about their awareness on RME treatment and oral hygiene maneuverers with scores from 0 (worst experience) to 10 (best experience).
Change in App questionnaire | Baseline (T0), 1 month (end of activations - T1), after 1.5 months (T2), after 3 (T3) and 6 months (T6)
  Parents and patients from Trial group will complete a questionnaire about Ortodontika application usefulness with scores from 0 (worst experience) to 10 (best experience).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding author.